CLINICAL TRIAL: NCT05398627
Title: Amygdala rtfMRI Neurofeedback for Borderline Personality Disorder
Brief Title: Neurofeedback for Borderline Personality Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kymberly Young (Other)
Collaborators: AE Foundation (Other)
Responsible Party: Sponsor-Investigator, Kymberly Young, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY22040107
Record Dates: First submitted 2022-05-25; First posted 2022-06-01 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Borderline Personality Disorder
Keywords: fMRI neurofeedback; amygdala
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Amygdala Neurofeedback (Experimental): Participants will undergo real-time fMRI neurofeedback training to increase their amygdala response while recalling positive autobiographical memories. 2 sessions will occur within a one week period.
  Interventions: Device: Amygdala Neurofeedback

INTERVENTIONS:
Device: Amygdala Neurofeedback — real-time feedback on the hemodynamic response of the amygdala during positive autobiographical memory recall

SUMMARY:
The goal of this study is to evaluate whether rtfMRI-nf training to increase the amygdala response to positive memories may serve as an intervention for borderline personality disorder.

DETAILED DESCRIPTION:
We will assess the treatment effects of real-time fMRI neurofeedback in adults with borderline personality disorder. This is an experimental longitudinal design where participants will be followed every two weeks after receiving 2 sessions of neurofeedback from the amygdala . Procedures involve a battery of self-report measures, fMRI and psychophysiological indices (heart rate, respiration).

ELIGIBILITY:
Inclusion Criteria:

* right-handed adults (ages 18 - 55) with a primary diagnosis of Borderline Personality Disorder according to diagnostic criteria in the Structured Interview for DSM Personality Disorders
* must be able to give written informed consent prior to participation
* unmedicated or stable on an SSRI antidepressant regime (at least 3 weeks to ensure symptoms are stable)
* English speaking

Exclusion Criteria:

* have a clinically significant or unstable cardiovascular, pulmonary, endocrine, neurological, gastrointestinal illness or unstable medical disorder
* Current moderate or severe DSM-V alcohol or substance use disorder, with the exception of nicotine or caffeine. Clinician will access subjects' alcohol and substance use on a case-by-case to determine whether specific cases of mild alcohol or substance use would also interfere with the effects of the intervention.
* have a history of traumatic brain injury
* are unable to complete MRI scan due to claustrophobia or general MRI exclusions (e.g., shrapnel inside body)
* are currently pregnant or breast feeding
* are unable to complete questionnaires written in English
* current (within 3 weeks of testing) use of any antipsychotics, benzodiazepines, beta-blockers, or other medications (except SSRI antidepressants) likely to influence cerebral blood flow. Effective medications will not be discontinued for the purposes of the study. Inclusion of patients on stable antidepressant medications was decided in order to allow generalization towards a real world population
* have a DSM-5 diagnosis of psychotic or organic mental disorder
* have any eye problems or difficulties in corrected vision.
* Serious suidicial ideation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Borderline Scale from the Personality Assessment Inventory at 12 weeks | Baseline vs 12 weeks
  Assessment of severity of borderline symptoms. This scale contains 24 items rated on a four-point scale (0=false to 3=very true). Scores range from 0-72, and are converted to T scores, with higher scores indicating more borderline symptoms. Scores below 59 indicate healthy, scores at or above 70T indicate the respondent is likely to have borderline personality disorder.

SECONDARY OUTCOMES:
Change from Baseline in Beck Depression Inventory at 12 weeks | Baseline vs 12 weeks
  Assessment of severity of depressive symptoms. This is a 21 item self-report scale with items rated from 0-3 and scores ranging from 0 to 63 with higher scores indicating worse depression. A score less than 13 is considered to be in the healthy range, scores 14-19 indicate mild depression, scores 20-28 indicate moderate depression, scores 29-63 indicate severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Kymberl Young, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made available to researchers who sign a data sharing agreement with the PI